CLINICAL TRIAL: NCT01119352
Title: A Phase 1, Single Centre, Single-Blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral AZD7687 After Administration of Multiple Ascending Doses in Overweight to Obese But Otherwise Healthy Male Subjects
Brief Title: AZD7687 Multiple Ascending Dose Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: D2710C00002; 2010-019112-21 (EudraCT Number)
Record Dates: First submitted 2010-05-06; First posted 2010-05-07 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Overweight; Obese
Keywords: Safety; tolerability; PK; healthy; overweight; obese
MeSH Terms: conditions — Overweight; Obesity | interventions — AZD7687

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD7687
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD7687 — Oral suspension, once daily. Starting dose of 1mg and with up to 4 dose escalations. Totally 8 doses.
  Arms: 1
Drug: Placebo — Oral suspension, once daily. Totally 8 doses
  Arms: 2

SUMMARY:
The aim of the study is to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of AZD7687 following multiple ascending dose administrations in in overweight to obese but otherwise healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures
* suitable veins for cannulation or repeated venepuncture.
* Have a body mass index (BMI) between 27 and 35 kg/m2

Exclusion Criteria:

* Fasting serum (S)-glucose ≥7.0 mmol/L or non-fasting S-glucose ≥11.1 mmol/L at screening.
* Any eating disorder or actively attempting to loose weight within 3 months prior to enrolment.
* Smoking more than 7 cigarettes per week from time of consent

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2010-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Safety variables (adverse events, vital signs, physical examination, telemetry, digital electrocardiograms (dECGs), safety 12-lead paper electrocardiograms (pECG), and clinical laboratory assessments) | Before, during and after dosing.

SECONDARY OUTCOMES:
Pharmacokinetics: Plasma and urine concentrations of AZD7687 and plasma and urine pharmacokinetic parameters | Information will be collected from the time of day -2 throughout the study.
Pharmacodynamic Biomarker sampling: (Triacylglycerol in serum, triacylglycerol, diacylglycerol, insulin and free fatty acids in plasma. Triacylglycerol and diacylglycerol in adipose tissue) | Information will be collected from the time of day -2 throughout the study.
Genetic: Blood sampling at one occasion during the study. | Once during study

CONTACTS AND LOCATIONS:
Overall Officials: Jan Eriksson, Study Director — AstraZeneca; Mirjana Kucajcic, Study Chair — AstraZeneca; Darren Wilbraham, Principal Investigator — Quintiles, Inc.
Locations (1):
- Research Site, London, United Kingdom